CLINICAL TRIAL: NCT01508325
Title: Comparison of Bisoprolol With Metoprolol Succinate Sustained-release on Heart Rate and Blood Pressure in Hypertensive Patients (CREATIVE Study)
Brief Title: Comparison of Bisoprolol With Metoprolol Succinate Sustained-release on Heart Rate and Blood Pressure in Hypertensive Patients
Acronym: CREATIVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Co., Ltd., China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EMR200006-520
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Results first posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-04

CONDITIONS: Hypertension
Keywords: Bisoprolol; Hypertension; Blood pressure; Heart rate
MeSH Terms: conditions — Hypertension | interventions — Bisoprolol; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bisoprolol (Experimental)
  Interventions: Drug: Bisoprolol
- Metoprolol (Active Comparator)
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: Bisoprolol — Subjects will receive bisoprolol fumarate (Concor®) at a dose of 5 milligram (mg) once daily orally as sustained release (SR) tablets for a period of 4 weeks. The dose of bisoprolol will be escalated to 7.5 mg orally once daily for next 4 weeks (Weeks 4 to 8) and to 10 mg orally once daily for the next 4 weeks (Weeks 8 to 12), if clinic systolic blood pressure (SBP) was greater than or equal to (>=) 140 millimeters of mercury (mmHg) and/or diastolic blood pressure (DBP) was >=90 mmHg measured every 4 weeks.
  Other Names: Concor
  Arms: Bisoprolol
Drug: Metoprolol — Subjects will receive metoprolol succinate (Betaloc SR) at a dose of 47.5 mg once daily orally as SR tablets for a period of 4 weeks. The dose of metoprolol will be escalated to 71.25 mg orally once daily for next 4 weeks (Weeks 4 to 8) and to 95 mg orally once daily for the next 4 weeks (Weeks 8 to 12) if clinic SBP was >=140 mmHg and/or DBP was >=90 mmHg measured every 4 weeks.
  Other Names: Betaloc SR
  Arms: Metoprolol

SUMMARY:
This is a multicentre, randomized, open-label parallel trial to demonstrate the superiority and/or non-inferiority of bisoprolol on metoprolol succinate sustained-release (SR) tablet in subjects with mild to moderate primary hypertension.

DETAILED DESCRIPTION:
Primary objectives:

To demonstrate that bisoprolol is superior in mean ambulatory heart rate and/or non-inferior in mean ambulatory DBP as compared with metoprolol SR in the last 4 hours after 12-week active treatment in subjects with mild to moderate essential hypertension (EH).

Secondary objectives:

1. To compare the efficacy of the 2 study drugs by 24h ambulatory monitoring by several parameters at different times (Example: blood pressure, heart rate, their variability, etc...) after 12-week treatment from baseline among subjects with mild to moderate EH
2. To evaluate safety of the two drugs
3. To evaluate the treatment compliance of the two drugs

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged: >=18 years and =<70 years old
2. EH who are suitable for mono-therapy, either mild to moderate EH patients who have not been treated with anti-hypertension drugs, or mild EH subjects who have taken anti-hypertension drug.
3. Clinic resting Heart Rate >=70 beats per minute (bpm)
4. Patients who have signed informed consent

Exclusion Criteria:

1. Subjects with contraindications according to the China Summary of Product Characteristics (SmPCs) of both bisoprolol and metoprolol SR, such as acute heart failure, second or third degree atrioventricular block (without a pacemaker), sick sinus syndrome, symptomatic bradycardia or symptomatic hypotension, severe bronchial asthma or severe chronic obstructive pulmonary disease, metabolic acidosis, etc.
2. Moderate EH patients who have used anti-hypertension drugs
3. Secondary hypertension
4. Subjects with history of coronary heart disease
5. Chronic or acute heart failure
6. Cerebrovascular events within 6 months before screening
7. Impaired hepatic or renal function (according to local lab standard)
8. Other protocol defined exclusion criteria could apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2011-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Serono Co., Ltd., China
Locations (1):
- Merck Serono Investigational Site, Changsha, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Bisoprolol: Subjects received bisoprolol fumarate (Concor®) at a dose of 5 milligram (mg) once daily orally as sustained release (SR) tablets for a period of 4 weeks. The dose of bisoprolol was escalated to 7.5 mg orally once daily for next 4 weeks (Weeks 4 to 8) and to 10 mg orally once daily for the next 4 weeks (Weeks 8 to 12), if clinic systolic blood pressure (SBP) was greater than or equal to (>=) 140 millimeters of mercury (mmHg) and/or diastolic blood pressure (DBP) was >=90 mmHg measured every 4 weeks.
- Metoprolol: Subjects received metoprolol succinate (Betaloc SR) at a dose of 47.5 mg once daily orally as SR tablets for a period of 4 weeks. The dose of metoprolol was escalated to 71.25 mg orally once daily for next 4 weeks (Weeks 4 to 8) and to 95 mg orally once daily for the next 4 weeks (Weeks 8 to 12) if clinic SBP was >=140 mmHg and/or DBP was >=90 mmHg measured every 4 weeks.
Period: Overall Study
Arm/Group | Bisoprolol | Metoprolol
Started | 93 | 93
Completed | 75 | 72
Not Completed | 18 | 21
Not completed — Withdrawal by Subject | 8 | 9
Not completed — Protocol Violation | 0 | 3
Not completed — Physician Decision | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 5 | 6
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) analysis population included all randomized subjects.
Groups:
- Bisoprolol: Subjects received bisoprolol fumarate (Concor®) at a dose of 5 mg once daily orally as SR tablets for a period of 4 weeks. The dose of bisoprolol was escalated to 7.5 mg orally once daily for next 4 weeks (Weeks 4 to 8) and to 10 mg orally once daily for the next 4 weeks (Weeks 8 to 12), if clinic SBP was >= 140 mmHg and/or DBP was >=90 mmHg measured every 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Bisoprolol | Metoprolol | Total
Number analyzed (Participants) | 93 | 93 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.10 (10.77) | 49.89 (10.46) | 50.49 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 56 | 92
  Male | 57 | 37 | 94

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Ambulatory Diastolic Blood Pressure (DBP) in the Last 4 Hours After 12-week Treatment
Description: Ambulatory blood pressure monitoring (ABPM) determined blood pressure 3 times hourly in the daytime and once hourly in the nighttime. Only monitoring data with valid data greater than or equal to (>=) 80 percent (%) was used for analysis. Each ABPM lasted for at least 24 hours. The first dynamic blood pressure monitoring was used as baseline. The difference between the mean ambulatory DBP observed in the last 4 hours after 12-week treatment and baseline was calculated to find out the change of mean ambulatory DBP at the end of the treatment.
Time Frame: Baseline and Week 12
Population: ITT analysis population included all the randomized subjects. 'n' signifies number of subjects evaluable for this outcome measure at given timepoints for each group, respectively
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol | Metoprolol
Number analyzed (Participants) | 93 | 93
mmHg
  Baseline (n=92, 93) | 85.28 (10.26) | 85.68 (11.59)
  Change at Week 12 (n=65, 66) | -4.45 (10.74) | -3.39 (11.23)

2. Primary Outcome: Change From Baseline in Mean Heart Rate in the Last 4 Hours After 12-week Treatment
Description: Pulse rate was measured by palpation on radial artery for 1 minute. Two measurements were made at least 1 to 2 minutes apart. Finally mean heart rate was recorded. The first measured heart rate was used as baseline heart rate. The difference between the last 4 hours heart rate after 12-week treatment and of the baseline heart rate was calculated to measure the change in mean heart rate at the end of the treatment.
Time Frame: Baseline and Week 12
Population: ITT analysis population included all randomized subjects. 'n' signifies number of subjects evaluable for this outcome measure at given timepoints for each group, respectively.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Bisoprolol | Metoprolol
Number analyzed (Participants) | 93 | 93
beats/min
  Baseline (n=92, 93) | 75.67 (10.58) | 73.99 (9.90)
  Change at Week 12 (n=65, 66) | -8.04 (12.65) | -4.75 (11.34)

3. Secondary Outcome: Change From Baseline in Mean Ambulatory Systolic Blood Pressure (SBP) in the Last 4 Hours After 12-week Treatment
Description: The ABPM determined blood pressure 3 times hourly in the daytime and once hourly in the nighttime. Only monitoring data with valid data >=80% was used for analysis. Each ABPM lasted for at least 24 hours. The first dynamic blood pressure monitoring was used as baseline. The difference between the mean ambulatory SBP observed in the last 4 hours after 12-week treatment and baseline was calculated to find out the change of mean ambulatory SBP at the end of the treatment.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol | Metoprolol
Number analyzed (Participants) | 93 | 93
mmHg
  Baseline (n=92, 93) | 132.68 (15.96) | 133.24 (16.69)
  Change at Week 12 (n=65, 66) | -5.97 (16.63) | -5.12 (15.12)

4. Secondary Outcome: Change From Baseline in Mean Ambulatory 24-hour Blood Pressure at Week 12
Description: The ABPM determined blood pressure 3 times hourly in the daytime and once hourly in the nighttime. Only monitoring data with valid data >=80% was used for analysis. Each ABPM lasted for at least 24 hours. The first dynamic blood pressure monitoring was used as baseline. The difference between the mean ABPM observed in the last 24 hours at Week 12 and baseline was calculated to find out the change of mean ABPM at the end of the treatment.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol | Metoprolol
Number analyzed (Participants) | 93 | 93
mmHg
  SBP: Baseline (n=92, 93) | 132.76 (12.88) | 135.43 (15.19)
  SBP: Change at Week 12 (n=68, 67) | -5.40 (14.59) | -4.54 (11.47)
  DBP: Baseline (n=92, 93) | 84.60 (8.22) | 86.94 (10.32)
  DBP: Change at Week 12 (n=68, 67) | -4.58 (9.01) | -3.78 (8.00)

5. Secondary Outcome: Change From Baseline in Mean Ambulatory Daytime Blood Pressure at Week 12
Description: The ABPM determined blood pressure 3 times hourly in the daytime. Only monitoring data with valid data >=80% was used for analysis. Each ABPM lasted for at least 24 hours. The first dynamic daytime blood pressure monitoring was used as baseline. The difference between the mean ambulatory daytime blood pressure observed at Week 12 and baseline was calculated to find out the change of mean ambulatory daytime blood pressure at the end of the treatment. Daytime in this study was defined as time between 06:00 am to 10:00 pm.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol | Metoprolol
Number analyzed (Participants) | 93 | 93
mmHg
  SBP: Baseline (n=92, 93) | 135.40 (13.11) | 138.31 (15.09)
  SBP: Change at Week 12 (n=68, 67) | -5.87 (15.29) | -5.16 (12.11)
  DBP: Baseline (n=92, 93) | 86.43 (8.88) | 88.86 (10.58)
  DBP: Change at Week 12 (n=68, 67) | -4.76 (9.34) | -3.82 (8.69)

6. Secondary Outcome: Change From Baseline in Mean Ambulatory Night-time Blood Pressure at Week 12
Description: The ABPM determined blood pressure once hourly in the nighttime. Only monitoring data with valid data >=80% was used for analysis. Each ABPM lasted for at least 24 hours. The first nighttime blood pressure monitoring was used as baseline. The difference between the mean ambulatory nighttime blood pressure observed at Week 12 and baseline was calculated to find out the change of mean ambulatory nighttime blood pressure at the end of the treatment. Nighttime in this study was defined as 10:00 pm to 06:00 am.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol | Metoprolol
Number analyzed (Participants) | 93 | 93
mmHg
  SBP: Baseline (n=92, 93) | 125.16 (14.14) | 127.15 (16.99)
  SBP: Change at Week 12 (n=68, 66) | -4.81 (14.31) | -2.65 (14.23)
  DBP: Baseline (n=92, 93) | 79.14 (7.68) | 81.19 (11.89)
  DBP: Change at Week 12 (n=68, 66) | -5.08 (9.29) | -3.39 (8.76)

7. Secondary Outcome: Change From Baseline in Mean Ambulatory Daytime Heart Rate at Week 12
Description: Pulse rate was measured by palpation on radial artery for 1 minute. Two measurements were made at least 1 to 2 minutes apart. Finally mean heart rate was recorded. The first measured daytime heart rate was used as baseline heart rate. The difference between the daytime heart rate at Week 12 treatment and of the baseline heart rate was calculated to measure the change of mean ambulatory daytime heart rate at the end of the treatment. Daytime in this study was defined as 06:00 am to 10:00 pm.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Bisoprolol | Metoprolol
Number analyzed (Participants) | 93 | 93
beats/min
  Baseline (n=92, 93) | 80.66 (8.85) | 78.94 (8.04)
  Change at Week 12 (n=66, 67) | -9.60 (10.76) | -3.85 (9.21)

8. Secondary Outcome: Change From Baseline in Mean Ambulatory Night-time Heart Rate at Week 12
Description: Pulse rate was measured by palpation on radial artery for 1 minute. Two measurements were made at least 1 to 2 minutes apart. Finally mean heart rate was recorded. The first measured heart rate was used as baseline heart rate. The difference between the nighttime heart rate at Week 12 treatment and of the baseline heart rate was calculated to measure the change of mean ambulatory nighttime heart rate at the end of the treatment. Nighttime was defined as 10:00 pm to 06:00 am.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Bisoprolol | Metoprolol
Number analyzed (Participants) | 93 | 93
beats/min
  Baseline (n=92, 93) | 67.73 (8.26) | 66.85 (7.38)
  Change at Week 12 (n=66, 66) | -4.72 (9.90) | -1.50 (7.24)

9. Secondary Outcome: Change From Baseline in 24-hour Blood Pressure Variability at Week 12
Description: The ABPM determined blood pressure 3 times hourly in the daytime and once hourly in the nighttime. Only monitoring data with valid data >=80% was used for analysis. Each ABPM lasted for at least 24 hours. The first dynamic blood pressure monitoring was used as baseline. The mean change in the blood pressure variability between the 24-hour blood pressure observed at Week 12 and baseline was calculated.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol | Metoprolol
Number analyzed (Participants) | 93 | 93
mmHg
  SBP variability: Baseline (n=91, 92) | 10.89 (3.45) | 10.45 (2.33)
  SBP variability: Change at Week 12 (n=66, 66) | -0.12 (3.56) | 0.09 (3.05)
  DBP variability: Baseline (n=91, 92) | 12.68 (3.63) | 12.09 (3.02)
  DBP variability: Change at Week 12 (n=66, 66) | 0.02 (3.54) | 0.76 (3.30)

10. Secondary Outcome: Blood Pressure Response Rate
Description: Blood pressure response was defined as DBP less than or equal to (=<) 90 mmHg or >=10 mmHg decrease in DBP from baseline. Blood pressure response rate was calculated as: number of subjects with blood pressure response divided by total number of subjects and multiplied by 100.
Time Frame: Week 12
Population: ITT analysis population included all randomized subjects. 'N' (number of subjects analyzed) signifies number of evaluable subjects for this outcome measure.
Measure: Number; unit: percentage of subjects
Arm/Group | Bisoprolol | Metoprolol
Number analyzed (Participants) | 75 | 72
percentage of subjects | 86.67 | 83.33

11. Secondary Outcome: Heart Rate Response Rate
Description: Heart rate response was defined as decrease in heart rate from baseline >=10 percent (%). Heart rate response rate was calculated by using the number of subjects with heart rate response divided by total number of subjects and multiplied by 100.
Time Frame: Week 12
Population: as for outcome 10
Measure: Number; unit: percentage of subjects
Arm/Group | Bisoprolol | Metoprolol
Number analyzed (Participants) | 75 | 72
percentage of subjects | 72.00 | 55.56

12. Secondary Outcome: Change From Baseline in Mean Ambulatory 24-hour Heart Rate at Week 12
Description: Pulse rate was measured by palpation on radial artery for 1 minute. Two measurements were made at least 1 to 2 minutes apart. Finally mean heart rate was recorded. The first measured heart rate was used as baseline heart rate. The difference between the last 24 hours heart rate at Week 12 and of the baseline heart rate was calculated.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Bisoprolol | Metoprolol
Number analyzed (Participants) | 93 | 93
beats/min
  Baseline (n=92, 93) | 77.45 (8.42) | 75.80 (7.53)
  Change at Week 12 (n=67, 67) | -8.46 (10.43) | -3.24 (8.03)

ADVERSE EVENTS:
Time Frame: From the first administration of the trial medication up to the end of the treatment (12 weeks)
Arm/Group | Bisoprolol | Metoprolol
Serious Adverse Events (participants affected / at risk) | 2/93 | 0/93
Other Adverse Events (participants affected / at risk) | 17/93 | 16/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bisoprolol (N=93) | Metoprolol (N=93)
Dizziness (Nervous system disorders) | 1 | 0
Transient attack (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bisoprolol (N=93) | Metoprolol (N=93)
Angina (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial ischemia (Cardiac disorders) | 0 | 1
Palpitation (Cardiac disorders) | 1 | 2
Ventricular premature contraction (Cardiac disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
High alanine aminotransferase (Investigations) | 1 | 0
High serum cholesterol level (Investigations) | 3 | 2
High blood glucose (Investigations) | 1 | 1
High blood triglycerides level (Investigations) | 2 | 4
High serum uric acid level (Investigations) | 0 | 2
Low high-density lipoprotein level (Investigations) | 1 | 0
High low-density lipoprotein level (Investigations) | 4 | 3
Urine leucocyte (positive) (Investigations) | 0 | 1
Urine protein (positive) (Investigations) | 1 | 0
Loss of appetite (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other